CLINICAL TRIAL: NCT03397602
Title: Exercise Training in Patients With Persistent or Permanent Atrial Fibrillation - a Multi-centre Randomized Controlled Trial
Brief Title: Exercise Training in Patients With Persistent or Permanent Atrial Fibrillation
Acronym: Exercise-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0906
Record Dates: First submitted 2018-01-04; First posted 2018-01-12 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; exercise
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity | interventions — Standard of Care; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard care (No Intervention): Participants do not participate in a on site structured exercise training program.
- standard care + MICE (Experimental): standard care + moderate-intensity continuous exercise training (MICE)
  Interventions: Behavioral: standard care + moderate-intensity continuous exercise training
- standard care + HIIT (Experimental): standard care + high-intensity interval training (HIIT)
  Interventions: Behavioral: standard care + high-intensity interval training

INTERVENTIONS:
Behavioral: standard care + moderate-intensity continuous exercise training — Participants will attend on-site moderate-intensity continuous exercise training two times weekly for 12 weeks.
  Arms: standard care + MICE
Behavioral: standard care + high-intensity interval training — Participants will attend on-site high-intensity interval training two times weekly for 12 weeks.
  Arms: standard care + HIIT

SUMMARY:
The main purpose of this project is to evaluate the effects of high-intensity interval training (HIIT) compared to moderate-intensity continuous exercise training (MICE) and standard care on exercise capacity and quality of life in patients with persistent or permanent atrial fibrillation. Positive findings are vitally important for these patients, given the condition's substantial morbidity, mortality and high economic costs.

DETAILED DESCRIPTION:
Recommended standards of care do not include the prescription of exercise to target and ameliorate the progressive health decline and overall feeling of well-being in patients with atrial fibrillation. Recent Standards for the Provision of Cardiac Rehabilitation of Ontario are calling for the consideration for referral and enrollment of patients with atrial fibrillation in cardiovascular rehabilitation - evidence is needed to support and confirm these efforts. The main purpose of this project is to evaluate the effects of high-intensity interval training (HIIT) compared to moderate-intensity continuous exercise training (MICE) and standard care on exercise capacity and quality of life in patients with persistent or permanent atrial fibrillation. Positive results from this study will identify a new intervention that: produces important improvements in patient-rated clinical, behavioural and exercise outcomes; provides mechanistic insight into the role of exercise training in the management of atrial fibrillation; requires minimal equipment; and, is appealing to patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. persistent or permanent atrial fibrillation;
2. rate controlled with a resting ventricular rate of equal to or less than 100 bpm;
3. able to perform a symptom-limited exercise test;
4. at least 40 years of age (i.e. participants must be 40 years or older);

Exclusion Criteria:

1. currently participating in routine exercise training (more than two times per week);
2. unstable angina;
3. diagnosed severe mitral or aortic stenosis;
4. diagnosed hypertrophic obstructive cardiomyopathy with significant obstruction;
5. pregnant, lactating or planning to become pregnant during the study period;
6. unable to provide written, informed consent, or
7. unwilling or unable to return for follow up at week 12.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2034-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life measured by the physical component summary (PCS) measure of the Short Form 36 Health Survey Questionnaire (SF-36). | baseline to 12 weeks
  Changes in quality of life measured by the physical component summary (PCS) measure of the Short Form 36 Health Survey Questionnaire (SF-36) from baseline to 12 weeks.
Changes in exercise capacity measured by VO2peak on a symptom-limited cardiopulmonary exercise test (CPET). | baseline to 12 weeks
  Changes in exercise capacity measured by VO2peak on a symptom-limited cardiopulmonary exercise test (CPET) from baseline to 12 weeks.

SECONDARY OUTCOMES:
Changes atrial fibrillation specific quality of life measured by the Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT). | baseline to 12 weeks
  Changes atrial fibrillation specific quality of life measured by the Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT). The AFEQT assesses 4 domains: symptoms, activities, treatment concern, treatment satisfaction, and a summary score that includes the first 3 domains. Patients will assess the impact of AF on their health status during the previous 4 weeks. Responses are presented as a 7-point Likert scale. Raw scores within each domain are transformed to a 0 (most severe symptoms) to 100 scale (no limitations or disability). The AFEQT is valid, reliable and sensitive to clinical change in patients with AF undergoing different therapeutic interventions.
Changes atrial fibrillation specific quality of life measured by the University of Toronto Atrial Fibrillation Severity Scale (AFSS). | baseline to 12 weeks
  Changes atrial fibrillation specific quality of life measured by the University of Toronto Atrial Fibrillation Severity Scale (AFSS) from baseline to 12 weeks. The AFSS is a disease-specific quality of life measure used to capture subjective and objective ratings of disease burden in patients with atrial fibrillation. It assesses atrial fibrillation burden (score 1-30; higher scores indicate higher burden); Global Well Being (a visual analogue scale ranging from 1-10, indicating a patient reports as having a worst possible life [0] to the best possible life[10]); AF symptom score (score of 0-35; higher scores indicate more bothered by AF symptoms); and health care utilization (score of 0-21; higher scores indicate greater health care utilization).
Changes in symptom burden measured by the Canadian Cardiovascular Society Severity of Atrial Fibrillation Scale. | baseline to 12 weeks
  Changes in symptom burden measured by the Canadian Cardiovascular Society Severity of Atrial Fibrillation Scale from baseline to 12 weeks.The CCS-SAF is a simple, concise, symptom-based severity scale to assess patient status. CCS-SAF scores range from 0 to 4, with highest values denoting severe impact of symptoms on quality of life and activities of daily living. The CCS-SAF has been validated in patients with atrial fibrillation.
Changes in quality of life measured by the mental component summary (MCS) measure of the Short Form 36 Health Survey Questionnaire (SF-36). | baseline to 12 weeks
  Changes in quality of life measured by the mental component summary (MCS) measure of the Short Form 36 Health Survey Questionnaire (SF-36) from baseline to 12 weeks. The SF-36 is a widely used and thoroughly validated, standardized, generic health survey with 36 questions. It yields an 8-scale (physical functioning; role-physical; bodily pain; general health; vitality; social functioning; role-emotional; and, mental health) profile of functional health and well-being scores as well as psychometrically-based physical (PCS) and mental (MCS) component summary scores.
Changes in heart rate control measured by 24-hour Holter ECG recordings and ECG recordings at each CPET. | baseline to 12 weeks
  Changes in heart rate control measured by 24-hour Holter ECG recordings and ECG recordings at each CPET from baseline to 12 weeks.
Changes in lower body muscular fitness measured by standard load tests. | baseline to 12 weeks
  Changes in lower body muscular fitness measured by standard load tests from baseline to 12 weeks.
Changes in volume and intensity of exercise measured directly by accelerometer. | baseline to 12 weeks
  Changes in volume and intensity of exercise measured directly by accelerometer from baseline to 12 weeks.
Changes in volume and intensity of exercise measured by self-report (exercise logs). | baseline to 12 weeks
  Changes in volume and intensity of exercise measured by self-report (exercise logs) from baseline to 12 weeks.
Changes in self-reported symptom frequency and severity measured by the 7-day symptom diary. | baseline to 12 weeks
  Changes in self-reported symptom frequency and severity measured by the 7-day symptom diary from baseline to 12 weeks.
Changes in self reported sleep patterns measured by the 7-day sleep diary. | baseline to 12 weeks
  Changes in self reported sleep patterns measured by the 7-day sleep diary from baseline to 12 weeks.
Changes in blood biomarker concentrations (participants at the University of Ottawa Heart Institute site only). | baseline to 12 weeks
  Changes in blood biomarker concentrations from baseline to 12 weeks (participants at the University of Ottawa Heart Institute site only).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - London Health Sciences Network, London, Ontario
  - University of Ottawa Heart Insititue, Ottawa, Ontario